CLINICAL TRIAL: NCT00774566
Title: A Comparison of Isolating the Pulmonary Veins With the Cryoballoon Catheter Versus Radiofrequency Segmental Isolation:a Randomized Controlled Prospective Non-inferiority Trial
Brief Title: PV-Isolation With the Cryoballoon Versus RF:a Randomized Controlled Prospective Non-inferiority Trial (FreezeAF)
Acronym: FreezeAF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Staedtisches Klinikum Karlsruhe (Other)
Collaborators: Heidelberg University (Other)
Responsible Party: Principal Investigator, Armin Luik, MD, Dr. Armin Luik, Staedtisches Klinikum Karlsruhe
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKK-001
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Results first posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Atrial Fibrillation
Keywords: catheter ablation; randomized; cryo; radiofrequency; atrial fibrillation; cryo-balloon; PV-Isolation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): segmental PVI using an irrigated tip catheter
  Interventions: Procedure: PV-Isolation RF
- 2 (Active Comparator): PVI using the Cryo-Balloon
  Interventions: Procedure: PV-Isolation Cryo

INTERVENTIONS:
Procedure: PV-Isolation RF — Radiofrequency
  Other Names: RF
  Arms: 1
Procedure: PV-Isolation Cryo — Cryo-Balloon
  Other Names: Cryo
  Arms: 2

SUMMARY:
This study is designed as a randomized, controlled, prospective, non-inferiority clinical trial, where the efficacy and safety of the cryoballoon ablation system (CE certificated) will be compared to the standard ablation technique (segmental isolation of the pulmonary veins) with radiofrequency energy. The primary study aim is to investigate whether the new cryoballoon ablation catheter system (Arctic Front CryoAblation Catheters, FlexCath Steerable Sheath, CryoCath Technologies Inc., Montreal, Canada) is at least as effective as radiofrequency (RF) segmental isolation in electrically disconnecting the pulmonary veins (PV) for the treatment of paroxysmal atrial fibrillation (AF) with respect to the absence of atrial arrhythmias without persistent complications after six and twelve months. Furthermore, the differences in terms of procedural complications such as pulmonary vein stenosis, phrenic nerve injuries, cerebrovascular accidents (CVA), pericardial tamponade, pain scores during the procedure, levels of cardiac inflammatory markers are compared between the treatment groups. The short and long-term clinical success as well as the costs of both systems will also be evaluated.

DETAILED DESCRIPTION:
Study objectives:

This study is designed as a randomized, controlled, prospective, non-inferiority clinical trial, where the efficacy and safety of the cryoballoon ablation system (CE certificated) will be compared to the standard ablation technique (segmental isolation of the pulmonary veins) with radiofrequency energy. The primary study aim is to investigate whether the new cryoballoon ablation catheter system (Arctic Front CryoAblation Catheters, FlexCath Steerable Sheath, CryoCath Technologies Inc., Montreal, Canada) is at least as effective as radiofrequency (RF) segmental isolation in electrically disconnecting the pulmonary veins (PV) for the treatment of paroxysmal atrial fibrillation (AF) with respect to the absence of atrial arrhythmias without persistent complications after six and twelve months. Furthermore, the differences in terms of procedural complications such as pulmonary vein stenosis, phrenic nerve injuries, cerebrovascular accidents (CVA), pericardial tamponade, pain scores during the procedure, levels of cardiac inflammatory markers are compared between the treatment groups. The short and long-term clinical success as well as the costs of both systems will also be evaluated.

Brief description of the cryoablation:

This catheter system uses nitrous oxide as refrigerant to cool the inside of the catheter tip or the balloon down to -30 to -70 degree in a closed system. Delivering the freezing energy on human cells for several minutes leads to their destruction. The destructed cells cannot conduct anymore. For PV isolation the cryoballoon can be placed at the orifice of the pulmonary veins to ablate the muscle connections between the PV- and left atrium (LA).

Study background:

AF is a common and disabling cardiac arrhythmia, affecting 600.000-700.000 persons in Germany. In addition to hemodynamic compromise and higher mortality rates, AF causes an increased risk of systemic emboli arising from the LA. The risk of stroke inpatients with nonvalvular AF is 5 to 7 times greater than in comparable patients without AF; overall, 20 - 25% of ischemic strokes are due to cardiac emboli, of which half arise in patients with nonvalvular AF. In addition to such proven mortality and morbidity risks, AF is associated with a substantial burden of symptoms, stemming from the arrhythmia itself, exacerbation of comorbid conditions such as congestive heart failure, associated anxiety over possible sequelae as well as the substantial burden of side effects from antiarrhythmic drugs (AAD). Currently available treatments are unsatisfactory for many reasons. AAD treatment has a relatively low efficacy even in patients suffering from paroxysmal AF, with frequent recurrences and a high incidence of intolerable drug side effects. Isolation of PVs using RF energy has shown considerable clinical success in the treatment of paroxysmal AF, but has been associated with serious complications, including PV stenosis, thromboembolic complications, cardiac perforation, phrenic nerve palsies, esophageal fistulae and pericardial tamponade. Furthermore, RF can be painful where as freezing with cryotherapy may be pain free.

CryoCath Technologies has developed and tested the Arctic Front™ Cardiac CryoAblation Catheter System (with the FlexCath™ Steerable Sheath) to allow the rapid formation of continuous cryoablation lesions at the PV ostia. Pre-clinical data have demonstrated long-term effectiveness of balloon cryoablation for permanent electrical isolation of the PVs with no risk of PV stenosis. Results from these pre-clinical studies suggest that no pulmonary venous stenosis and no thromboembolic incidents have occurred even with multiple 4 or 8-minute cryoenergy deliveries. However, achieving an adequate therapeutic effect using focal or linear cryolesions often required multiple applications and lengthy procedure times. Balloon cryoablation of subjects with PAF has been studied in PS-011, a feasibility study of the Arctic Front™ Balloon Cardiac CryoAblation Catheter System, in conjunction with the Freezor® MAX and Xtra and the Arctic Circler Linear™ Cardiac CryoAblation Catheter. Twenty (20) subjects were enrolled at two European centers using the 23 mm Arctic Front™ Balloon, and an additional 7 subjects were enrolled using 28 mm Arctic Front™ Balloon. Acute procedural success was 100%, and long term follow-up reveals a high rate of freedom from recurrent AF. A low incidence of adverse events was noted, with two patients experiencing reversible loss of phrenic nerve capture during the procedure. Both patients recovered fully. Of the original 20 subjects treated with the 23 mm balloon, 16 / 20 (80%) were AF-free between the 6 and 12 month follow-up visits. Of the additional 7 subjects treated with the 28 mm balloon, 5 / 6 (83%) were AF free through 6 months. Another non-randomized feasibility study of the Arctic Front™ 23 mm Balloon Cardiac CryoAblation Catheter System under protocol PS-012 has completed enrollment at four centers in the United States. Based on incompletely monitored data, as of July 12th, 2006, 31 patients have undergone a successful cryoablation procedure with Acute Procedural Success (isolation of ≥ 3 PVs) in 100% (31 / 31 subjects). Electrical isolation was achieved in 129 / 130 PVs (99.3%). A total of 67 adverse events (AE) have been reported, and no deaths. Nine (9) serious AEs have been reported. Four device related serious AEs involved changes in phrenic nerve conduction: 3 patients had cryoablation discontinued immediately and nerve function recovered completely by 1 month, and the fourth subject had transient loss of capture during the procedure, followed at the 1 month visit by shortness of breath, a viral infection and slight paralysis of a hemidiaphragm. Two other device related serious AEs were a pericardial tamponade requiring pericardiocentesis and hospitalization, and a right groin hematoma. Three additional non-device related serious AEs included one episode of chest pain, one instance of right neck bleeding after vascular access and one instance of left groin site bleeding after vascular access. Long term follow-up for PS-012 is incomplete, but 17 subjects have reached 3 months, and 14 / 17 (82%) are free from recurrent AF. Only one of these 14 subjects was on a previously failed AF drug, giving a 76% (13 / 17) rate of freedom from recurrent AF off drugs.

Additional data from another non-randomized clinical study are now available (Neumann et al. Circumferential pulmonary vein isolation with the cryoballoon technique. JACC 2008, Vol 52(4); 273-8). 346 patients consecutive patients in three German centers have undergone a successful cryoablation therapy. The study population consisted of 293 patients with paroxysmal and 53 patients with persistent atrial fibrillation. Isolation of the pulmonary veins was achieved in 97% where as freedom from documented paroxysmal atrial fibrillation was achieved in 74% after a median follow-up of 12 month. No death and no PV narrowing occurred. In 26 patients (7,5%) a phrenic nerve palsy could be observed. The majority of the patients recovered within 6 month, all patients recovered within 12 month.

Based on these encouraging results this randomized clinical study has been designed to provide valid scientific evidence of the safety and effectiveness of the Arctic Front™ Cardiac CryoAblation Catheter System (with a FlexCath™ Steerable Sheath) to electrically isolate PVs in patients with PAF by comparing it with segmental isolation with RF-energy, which represents the most widely accepted and used energy form in AF-ablation procedures. Compared to the RF ablation procedures PV isolation with the Cryo Balloon technique is easier and faster to perform and there is no need for expensive additional mapping systems to avoid current dreaded complications such as PV-stenosis or esophageal fistula.

Eligibility criteria:

Inclusion criteria:

* Documented paroxysmal PAF: PAF diagnosis, 2 episodes of PAF within the last 3 months, at least 1 episode of PAF must be documented.
* Age 18-75
* Documented effectiveness failure of at least 1 AAD including beta-blockers

Exclusion criteria:

* AAD usage < 3 half life periods (except beta-blocker)
* LA size > 55 mm
* LA thrombus
* Previous LA ablation/surgery, structural heart disease, heart failure class III-IV
* Hypertrophic cardiomyopathy
* Mitral prosthesis
* Unstable angina
* Uncontrolled hyperthyroidism
* Stroke or TIA within 6 months
* Myocardial infarction within 2 months
* Cardiac surgery within 3 months
* Thrombocytosis, thrombocytopenia
* Any condition contraindicating chronic anticoagulation
* EF <40%
* Pregnancy
* Life expectancy <1year

Preprocedural investigations:

* Transesophageal echocardiography to exclude LA thrombus in each patient before each ablation
* CT or MRT of the LA (optional)

Ablation procedure:

After venous and arterial access a single or double transseptal puncture is performed. In both groups a pulmonary vein angiography must be performed before and after PV - isolation for all of the PVs. PV - potentials must be recorded before and after PV - isolation with a circular mapping catheter. In group 1, the RF - ablation procedure is performed using an open 4 mm irrigated tip catheter in combination with a 3D - navigation system. It is recommended, that the 3D - navigation system should be able to display all mapping and ablation catheters. An antral PV - isolation will be performed. In group 2 a cryoablation of the PV - ostia using either the 28 mm or the 23 mm cryo-balloon will be attempted. At least two cryoenergy applications of 300 - 360 sec must be performed in each PV. Additional cryoenergy applications can be delivered if necessary to achieve complete isolation. The 28 mm cryoballoon should be used preferentially for all veins. If a complete isolation could not be achieved with the 28 mm cryoballoon ablation, a switch over to the 23 mm balloon is possible; otherwise touch-ups with a conventional cryocatheter (Freezor® Max, CryoCath) will be performed.

In both groups the aim is to completely isolate the PVs. The upper limit of RF - or cryo - applications is dependent on the procedure duration and the clinical condition at the time of the procedure and left to the physician´s decision. After the ablation all the pulmonary veins should be assessed with angiography to detect an ablation mediated PV - stenosis.

Anticoagulation: All patients should be anticoagulated four weeks before and at least six months after the index procedure. During the procedure the activated clotting time (ACT) must be kept between 250-350 sec by i.v. heparin administration.

AAD: All AAD should be discontinued 4 to 5 half-life periods before the procedure. No AAD will be prescribed (except betablocker) after the procedure.

Follow-up:

All patients will be monitored during the hospital stay after the procedure (the first 24-48h). Additional clinical visits will be performed at three, six, nine and twelve months after the last procedure. Another MRI or CT scan should be performed at the third month to re-evaluate the PVs and at least one 24h holter ECG recording to screen for symptomatic or asymptomatic atrial arrhythmias (AF, AT) has to be done. An event recorder or holter ECG to reveal the long-term recurrences will be given at the six and twelve month follow-up (for minimum of seven days, preferably 14 days) 22. In case of a recurrence a second procedure can be performed six months after the index procedure. The procedure of choice for the recurrences will be the same modality to which the patient originally had been randomized

Endpoints:

Primary endpoints:

Combined endpoint out of:

Absence of atrial arrhythmias and absence of persistent complications six and twelve months after the procedure .

Secondary endpoints:

Short- and mid-term clinical success Long-term clinical success Total radiation exposure Total procedure duration Pain sensation during the procedure Quality of life Changes in cardiac markers (CK, troponin, CRP) Bleedings Costs

Biometrical concept:

Randomization The randomization numbers will be allocated to the two groups in balanced permuted blocks using the random number generator of the validated software SAS®. To avoid any potential of predicting the group allocation of future patients, the block length is fixed in a separate document that is withheld from the study site. Sealed envelopes are produced labeled with the randomization number. Inside of the sealed envelope, a data sheet defines the group allocation of the patient with the respective randomization number. On enrollment in the study, each patient receives the randomization envelope in consecutive order of inclusion in the study. Basic characteristics of the patient and day of randomization are documented on the data sheet in order to allow a check whether the randomization scheme was observed strictly.

Statistical considerations:

Test problem and analysis of primary endpoint The primary objective of this trial is to demonstrate non-inferiority of isolating PVs procedure with the cryoballoon catheter (CC) as compared to radiofrequency isolation (RF) with respect to the primary endpoints "absence of atrial arrhythmias and absence of persistent complications six and twelve months after the procedure", respectively. For this purpose, the following test problems will be assessed: Null hypothesis H0: pCC (rate of absence of atrial arrhythmias and absence of persistent complications twelve months after the procedure with CC) - pRF (rate of absence of atrial arrhythmias and absence of persistent complications twelve months after the procedure with RF) -d versus alternative hypothesis H1: pCC - pRF > -d, where d = 0.15 defines the non-inferiority margin that is deemed to be acceptable in view of the advantages of CC with respect to aspects other than the primary endpoint. The analogous test problem is formulated for the endpoint after six months follow up. These test problems will be analyzed applying the non-inferiority test for rates according to Farrington and Manning17 at a one-sided significance level of a = 2.5%. The following multiple test procedure for hierarchically ordered hypotheses is applied to account for the multiplicity in primary endpoints: The null hypothesis formulated for the six months outcome is only tested if the null hypothesis for the twelve months outcome can be rejected; otherwise both null hypotheses are accepted. If both null hypotheses can be rejected, the null hypotheses H0g are tested at one-sided level a = 2.5% for margins g < d as long as H0g has to be accepted for a value gSTOP. Then, non-inferiority of CC as compared to RF has been shown for all non-inferiority margins g < gSTOP. This multiple test procedure controls the overall type I error rate a18, 19.

Confirmatory analysis will be primarily based on the FAS which is consistent with the intention-to-treat (ITT) principle by including all patients who were randomized to the two groups. This approach reflects the idea that the study should match as close as possible to the conditions in clinical practice. However, the PP analysis plays an important role particularly in non-inferiority studies, and therefore the results of the PP analysis set are to be interpreted and discussed with special attention in parallel to the ITT analysis.

Determination of the sample size Sample size calculation is based on the following considerations. In view of the advantages of CC as compared to RF in dimensions other than the primary endpoints, an inferiority by a difference in rates of 0.15 for CC as compared to RF with respect to the two primary outcomes is deemed to be acceptable. Therefore, the non-inferiority range was set equal to d = 0.15. On the basis of previous studies and experiences with the procedures16, equal rates of pCC = pRF = 0.78 are assumed for sample size calculation. Under these assumptions, the sample size required to achieve a power of 1 - b = 80% for the one-sided Farrington-Manning test at level a = 2.5% amounts to 2 x 122 = 244 patients17. In order to cope with the uncertainty about the assumed overall rate of 0.78, a sample size review is performed after 150 patients are randomized or the outcome of the primary variable is available for 100 patients, respectively, depending on which of the events occurs first. No significance test is performed then and hence there is no option for early stopping with rejection of the null hypothesis. Instead, the overall rate for the primary variable is estimated based on the available data and the sample size is recalculated employing the obtained value in the sample size formula (i.e. pCC = pRF = estimated overall rate) and leaving the values for a, 1-b, and d as above. It was shown that this procedure does not affect the type I error rate of the analysis20.

Each patient's allocation to the different analysis populations (full analysis set (FAS) according to the intention-to-treat (ITT) principle, per protocol (PP) analysis set, safety analysis set) will be defined prior to the analysis. The allocation will be documented in the statistical analysis plan.

During the data review before start of any analysis, deviations from the protocol will be assessed as "minor" or "major". Major deviations from the protocol will lead to the exclusion of a patient from the PP analysis set. If a patient discontinues from the study prematurely, missing data with respect to the primary outcome variable will be replaced by ICA-r method19.

Analysis of secondary endpoints The secondary variables will be analyzed descriptively by tabulation of the measures of the empirical distributions. According to the scale level of the variables, means, standard deviations, median, 1st and 3rd quartiles as well as minimum and maximum or absolute and relative frequencies, respectively, will be reported. Logistic regression models will be applied to assess the effects of potential risk factors on primary and secondary efficacy variables. Additionally, for variables with longitudinal measurements the time courses of individual patients and summarized by treatment groups will be compared. Descriptive p-values of the corresponding statistical tests comparing the treatment groups and associated 95% confidence intervals will be given.

The safety analysis will be based on the set of all patients for which one of the procedures was applied. Adverse and serious adverse events as well as complications will be tabulated, absolute and relative frequencies; the severity and the relationship to the procedure will be given and compared between the groups. Cardiac markers will be described and interpreted with respect to the reference values, and the measures describing the empirical distributions of the changes are calculated. Additionally, for each cardiac marker, shift tables presenting changes between the categories "normal" and "abnormal" will be given per treatment group.

Definitions:

Acute procedural success: Successfully isolation of all the pulmonary veins

Clinical success:

Absence of any atrial arrhythmias sustaining longer than 30 seconds evaluated either by telemetric monitoring, 24 hour ECG recordings or event recorder Short-term clinical success: from the procedure until hospital discharge Mid term clinical success: up to three months after the procedure Long-term clinical success: up to six months after the procedure

Procedure related complications: Any new PV-stenosis, phrenic nerve palsy, CVA, bleedings or vascular complications which occurs during and/or within 48 hours after the procedure.

Persistent complications:

Any procedure related complication lasting longer than 6 months after the procedure and either classified as major complication or still symptomatic.

PV-stenosis:

Angiographic late lumen loss of any PV in comparison to the pre-procedural data Minor: asymptomatic or stenosis less than 50%; Major: symptomatic or stenosis greater than 50%. 3 months after the procedure either a computer tomography, magnet resonance tomography or a echocardiography will be performed to re-evaluate the severity grade of the stenosis. If a stenosis is detected a repeat diagnosis will be performed at 6 month.

Phrenic nerve palsy:

Radiological restricted movement of the diaphragm Minor: asymptomatic or less than 50% restriction Major: symptomatic or more than 50% restriction In cases of persistent symptoms due to phrenic nerve palsy at least one fluoroscopy will be performed up to the 6 months follow-up to verify the restriction of the diaphragm.

Bleedings and vascular complications:

Minor: Any bleeding or vascular complication (hematoma, pseudoaneurysm, atriovenous fistula) requiring prolonged hospitalization but could be managed conservatively Major: Any bleeding or vascular complication requiring additional therapy (i.e. surgery, transfusion therapy)

CVA: Every new TIA or stroke after the procedure.

Quality of life:

Before and at every clinical visit patients will be ask to complete a standardized questionnaire to evaluate the symptomatic and life restrictiveness originating from the arrhythmia.

Pain After venous and arterial puncture and after the complete procedure the patients will be asked to grade their sensation of pain (range 1-10)

Costs Standard prices for consumable material such as catheters, electrodes, refrigerant per EP study will be evaluated. Purchase or leasing prices i.e. for a mapping system or the cryo console will not be considered.

Abbreviations:

AAD: Antiarrhythmic drugs AE: Adverse events AF: Atrial fibrillation AT: Atrial tachycardia CVA: Cerebrovascular accident EF: Ejection fraction LA: Left atrium PAF: Paroxysmal atrial fibrillation PNP: Phrenic nerve palsy PV: Pulmonary vein RF: Radiofrequency energy TIA: Transient ischemic attack

ELIGIBILITY:
Inclusion Criteria:

* Documented paroxysmal PAF: PAF diagnosis, 2 episodes of PAF within the last 3 months, at least 1 episode of PAF must be documented.
* Age 18-75
* Documented effectiveness failure of at least 1 AAD including beta-blockers

Exclusion Criteria:

* AAD usage < 3 half life periods (except beta-blocker)
* LA size > 55 mm
* LA thrombus
* Previous LA ablation/surgery, structural heart disease, heart failure class III-IV
* Hypertrophic cardiomyopathy
* Mitral prosthesis
* Unstable angina
* Uncontrolled hyperthyroidism
* Stroke or TIA within 6 months
* Myocardial infarction within 2 months
* Cardiac surgery within 3 months
* Thrombocytosis, thrombocytopenia
* Any condition contraindicating chronic anticoagulation
* EF < 40%
* Pregnancy
* Life expectancy < 1 year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2008-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claus Schmitt, MD, Study Chair — Staedtisches Klinikum Karlsruhe; Armin Luik, MD, Principal Investigator — Staedtisches Klinikum Karlsruhe
Locations (1):
- Staedtisches Klinikum, Karlsruhe, Baden-Wurttemberg, Germany

REFERENCES:
- [Result] Neumann T, Vogt J, Schumacher B, Dorszewski A, Kuniss M, Neuser H, Kurzidim K, Berkowitsch A, Koller M, Heintze J, Scholz U, Wetzel U, Schneider MA, Horstkotte D, Hamm CW, Pitschner HF. Circumferential pulmonary vein isolation with the cryoballoon technique results from a prospective 3-center study. J Am Coll Cardiol. 2008 Jul 22;52(4):273-8. doi: 10.1016/j.jacc.2008.04.021. PMID 18634982
- [Derived] Luik A, Kunzmann K, Hormann P, Schmidt K, Radzewitz A, Bramlage P, Schenk T, Schymik G, Merkel M, Kieser M, Schmitt C. Cryoballoon vs. open irrigated radiofrequency ablation for paroxysmal atrial fibrillation: long-term FreezeAF outcomes. BMC Cardiovasc Disord. 2017 May 25;17(1):135. doi: 10.1186/s12872-017-0566-6. PMID 28545407

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 322 patients were included, with 7 not receiving treatment as part of the trial because of a withdrawal of consent but without knowing group assignment leaving 315 patients randomly assigned. This resulted in a final ITT population of 315 patients.
Groups:
- Radiofrequency (RF) Ablation: Patients in this arm were treated with the established RF ablation approach with an open irrigated tip ablation catheter for the treatment of paroxysmal atrial fibrillation. All patients have at least experienced 2 episodes of AF within the last 3 month before inclusion.
- Cryo Balloon(CB) Ablation: Patients in this arm were treated with the cryo balloon ablation technique for the tretment of paoxysmal atrial fibrillation (AF). All patients have at least experienced 2 episodes of AF within the last 3 month before inclusion.
Period: Overall Study
Arm/Group | Radiofrequency (RF) Ablation | Cryo Balloon(CB) Ablation
Started | 159 | 156
6 Month Follow up | 154 | 150
12 Month Follow up | 141 | 141
Completed | 141 | 141
Not Completed | 18 | 15
Not completed — Protocol Violation | 18 | 15

BASELINE CHARACTERISTICS:
Groups:
- RF Ablation: Patients that have been randomized into the RF ablation group and have recieved the treatment as per protocol
- CB Ablation: Patients that have been randomized into the cryo balloon ablation group and have recieved the treatment as per protocol
- Total: Total of all reporting groups
Arm/Group | RF Ablation | CB Ablation | Total
Number analyzed (Participants) | 159 | 156 | 315
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [54 to 67] | 61 [54 to 66] | 61 [54 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 56 | 124
  Male | 91 | 100 | 191
Diabetes mellitus [Count of Participants; unit: Participants] | 17 | 14 | 31
Hypertension [Count of Participants; unit: Participants] | 103 | 96 | 199
Stroke [Count of Participants; unit: Participants] — patients with a previous history of Stroke
  Participants | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Combined Endpoint Out of: Absence of Atrial Arrhythmias and Absence of Persistent Complications at Six Months After the Index Procedure
Description: Redo procedures were only allowed after the 6 month follow up. Redo procedures had to be performed using the same energy source. No ADD administration was allowed after the ablation procedure.
Time Frame: Six months after procedure
Measure: Count of Participants; unit: Participants
Groups:
- RF Ablation: patients that have undergone RF ablation
- CB Ablation: patients that have undergone CB ablation
Arm/Group | RF Ablation | CB Ablation
Number analyzed (Participants) | 154 | 150
Participants | 99 | 98

2. Primary Outcome: Combined Endpoint Out of: Absence of Atrial Arrhythmias and Absence of Persistent Complications Twelve Months After Procedure.
Description: Including redo procedures. Redo procedures were only allowed after the 6 month follow up. Redo procedures had to be performed using the same energy source. No ADD administration was allowed after the ablation procedure.
Time Frame: Twelve month after the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | RF Ablation | CB Ablation
Number analyzed (Participants) | 141 | 141
Participants | 103 | 105

3. Secondary Outcome: Long-term Clinical Success
Description: Absence of atrial arrhythmias at twelve months after procedure.
Time Frame: Twelve month after the procedure
Population: patients that meet all protocol criteria (PP) after 12 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | RF Ablation | CB Ablation
Number analyzed (Participants) | 159 | 156
Participants | 141 | 141

4. Secondary Outcome: Total Radiation Exposure
Description: Analyzes the differences in x-ray dosage exposure during the procedures
Time Frame: at time of the procedure
Population: all patients the have been treated per protocol (PP)
Measure: Median (Inter-Quartile Range); unit: cGy
Arm/Group | RF Ablation | CB Ablation
Number analyzed (Participants) | 159 | 156
cGy | 50.0 [24.0 to 79.0] | 61.5 [36.0 to 97.0]

5. Secondary Outcome: Total Procedure Duration
Description: Analyzes the differences in procedure duration
Time Frame: at time of the procedure
Population: all patients that have been treated per protocol (PP)
Measure: Median (Inter-Quartile Range); unit: min
Arm/Group | RF Ablation | CB Ablation
Number analyzed (Participants) | 159 | 156
min | 162.0 [133.0 to 200.0] | 151.0 [119.0 to 182.0]

6. Secondary Outcome: Major Adverse Events
Description: calculated as freedom from any major adverse events until 12 month follow up period
Time Frame: procedure date till 12 month after the procedure
Population: all patients that have been treated per protocol (PP)
Measure: Count of Participants; unit: Participants
Arm/Group | RF Ablation | CB Ablation
Number analyzed (Participants) | 159 | 156
Participants
  patietns without any event | 147 | 144
  patients with missing information | 12 | 12

7. Secondary Outcome: Mid-term Clinical Success
Description: Absence of atrial arrhythmias at six months after procedure.
Time Frame: Six month after the procedure
Population: patients that meet all protocol criteria (PP) after 6 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | RF Ablation | CB Ablation
Number analyzed (Participants) | 159 | 156
Participants | 154 | 150

ADVERSE EVENTS:
Time Frame: at procedure, 6 and 12 month after procedure
Groups:
- RF Ablation: all patients that underwent RF ablation procedure
- CB Ablation: all patients that underwent CB ablation procedure
Arm/Group | RF Ablation | CB Ablation
All-Cause Mortality (participants affected / at risk) | 0/159 | 0/156
Serious Adverse Events (participants affected / at risk) | 4/159 | 9/156
Other Adverse Events (participants affected / at risk) | 3/159 | 8/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RF Ablation (N=159) | CB Ablation (N=156)
Vascular complication (Vascular disorders) | 4 (4) | 5 (5) — Any bleeding or vascular complication requiring additional therapy
Phrenic nerve palsy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — Radiological restricted movement of the diaphragm. symptomatic or more than 50% restriction
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2) — needed treatment (puncture, surgery) and prolonged hospital stay
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RF Ablation (N=159) | CB Ablation (N=156)
Valscular complication (Vascular disorders) | 1 (1) | 2 (2) — Any bleeding or vascular complication requiring prolonged hospitalization but could be managed conservatively
Phrenic nerve palsy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6) — Radiological restricted movement of the diaphragm. asymptomatic or less than 50% restriction
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0) — no prolongation of hospital stay, treated conservatively

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This is an investigator initiated study. The study was supported with 20.000 EUR to acquire Holter monitor devices by CryoCath/Medtronic.